CLINICAL TRIAL: NCT00492414
Title: Costs of Lost Productive Time Among Korean Workers With Panic Disorder and Effect of Treatment With Paroxetine Controlled Release
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: COL110010
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2007-08-08 (Estimated); Status verified 2007-03

CONDITIONS: Panic Disorder
Keywords: Panic disorder (PD)
MeSH Terms: conditions — Panic Disorder

INTERVENTIONS:
Drug: Paroxetine CR

SUMMARY:
Panic disorder(PD)is a disabling psychiatric condition associated with significant impairment in psychosocial, occupational functioning and quality of life, as mentioned by mogotsi et al. So, most patients with panic disorder suffers from the consequences of the impairment in occupational function. This impairment is not only individual problem, but also social one. Since productivity is very important item required to employees, lost productive time among workers with psychiatric illness should be reduced by the proper management. But few data were reported in this field by now.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients aged 20-50 years
2. In female, is eligible to enter this study if she is if

   * Non-childbearing potential(note:women who are 6 months post-menopausal are not considered women of child-bearing potential)
   * child-bearing potential, has a negative urine dipstick pregnancy test, and is practicing a clinically acceptable method of contraception such as oral contraception, surgical sterilization, I.U.D.,systemic contraception, or double barrier contraception(any two of diaphragm/spermicidal foar/condom)
3. Subject currently meets the diagnosis for PD according to korean version of Anxiety Disorder Interview Schedule for DSM-IV(ADIS-IV) through a comprehensive psychiatric evaluation and not being treated currently.
4. Subject must have the ability to comprehend the key components of the consent form and provide informed consent.

Exclusion Criteria:

1. Subject who has a history of any other major medical or psychiatric illnesses except PD or PD with major depressive disorder.
2. Subject who retired or left his job or who plan to retire within two years.
3. is a current homicidal or suicidal risk in the investigator's judgement.
4. is currently pregnant, lactating or planning to become pregnant within the next 3 months
5. is currently participating in any other clinical trial or taking any non-approved or experimental medication.

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Min Woo, Master, Principal Investigator — Seoul Paik Hospital, Inje University
Locations (1):
- Seoul Paik Hospital, Inje University, Seoul, Seoul, South Korea